CLINICAL TRIAL: NCT06901297
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial of the Efficacy and Safety of Raphamin in the Treatment of Acute Rhinosinusitis in Adult Patients
Brief Title: The Efficacy and Safety of Raphamin in the Treatment of Acute Rhinosinusitis in Adult Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-011
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Rhinosinusitis; Rhinosinusitis Acute
Keywords: Rhinosinusitis; Acute
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Per os without food. The tablet should be kept in mouth until completely dissolved.
  On day 1 of treatment, 8 tablets should be taken using the following regimen: 1 tablet every 30 minutes for the first 2 hours (5 tablets in total for 2 hours), then 1 more tablet 3 times at equal intervals during the same day. On day 2 and onwards, 1 tablet should be taken 3 times a day. The duration of treatment is 5 days.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Placebo using the Raphamin dosage regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Oral administration
  Other Names: MMH-407
  Arms: Raphamin
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
Multicenter double-blind placebo-controlled randomized in parallel groups clinical trial of the efficacy and safety of Raphamin in the treatment of acute rhinosinusitis in adult patients.

DETAILED DESCRIPTION:
A multicenter, double-blind, placebo-controlled, randomized, parallel-group clinical trial.

The trial will enroll outpatients of either gender aged 18 to 75 years with clinical manifestations of acute rhinosinusitis (ARS) within the first 48 hours after the disease onset. Patient recruitment will be conducted during the seasonal incidence of acute respiratory viral infection (ARVI). After the patient signs the information sheet and informed consent form for participation in the clinical trial, the medical history will be collected, thermometry, objective examination, laboratory tests will be performed, concomitant diseases and concomitant therapy will be recorded. The severity of ARS symptoms will be assessed using Major Symptom Score (MSS). Initially (Day 1) and on Visits 2 (Day 4) and 3 (Day 7), the patient together with the investigator, fills in the MSS scale and completes the Sino-Nasal Outcome Test questionnaire for assessing the quality of life of patients with diseases of the nose and paranasal sinuses (SNOT-22).

If all inclusion criteria are met and there no any exclusion criteria, at Visit 1 (Day 1), the patient is randomized into one of two groups: Group 1 patients will receive Raphamin according to the dosage regimen for 5 days; Group 2 patients will receive Placebo using the Raphamin dosage regimen for 5 days.

The trial uses an electronic patient diary (EPD) where the patient daily morning and evening will make records axillary body temperature (measured with a classic mercury-free thermometer) and symptoms of the disease (according to the MSS). In addition, administration of basic therapy drugs (if applicable) as well as any possible worsening of the patient's condition (if applicable, to assess safety / to record adverse events) should also be recorded in the patient diary. The investigator will instruct the patient on how to complete the diary. At Visit 1, the patient will record the severity of ARS symptoms and body temperature in the diary together with the physician.

The patient will be observed for 14 days (screening, randomization - up to 1 day, treatment - 5 days, follow-up - up to 14 days).

During the treatment and follow-up period, patients/physicians will pay 3 visits, on days 1, 4 and 7 (Visits 1, 2 and 3) - at a medical center or at home; a phone visit (Visit 4) will be on day 14.

At Visits 2 and 3, the investigator performs objective examination, records changes in the disease symptoms, concomitant therapy, and controls the filling of the diary, evaluates the patient's compliance (Visit 3). At Visit 4 (a phone visit), the investigator evaluates safety, collects information about the patient's condition, the presence/absence of complications, the use of antibiotics, and the presence/absence of hospitalization of the patient.

Symptomatic therapy and therapy for concomitant diseases will be permitted during the trial except for the drugs listed under "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 - 75 years.
2. Diagnosis of acute rhinosinusitis:

   * 8-12 points on MSS scale;
   * no more than 3 severe symptoms (3 points on the MSS scale)
   * facial pain/heaviness in the facial area 1-2 points on the MSS scale.
3. Disease duration up to 48 hours (from the onset of the first symptoms of the disease).
4. Availability of a patient information sheet and an informed consent form for participation in the clinical trial signed by the patient.
5. Patients who agreed to use a reliable method of contraception during the study (for men and women of reproductive potential).

Exclusion Criteria:

1. Symptoms of acute bacterial rhinosinusitis (three or more of those below):

   * fever of ≥ 38.0°C;
   * the second wave of ARS symptoms;
   * one-sided process;
   * facial pain/pressure of 3 points (on the MSS scale).
2. Recurrent ARS (≥4 episodes of ARS per year with complete resolution of symptoms between episodes).
3. Odontogenic rhinosinusitis.
4. Allergic (seasonal or year-round) rhinitis.
5. Nasal polyps or clinically significant nasal septum deviation.
6. Concomitant otitis.
7. Use of intranasal or systemic corticosteroids for 30 days prior to the screening visit.
8. Use of intranasal or systemic antibiotics for 30 days prior to the screening visit.
9. Surgery for the nasal cavity and paranasal sinuses during the last 6 months before the screening visit.
10. Any other surgery during the last 3 months.
11. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
12. Suspected bacterial infection of any localization requiring the administration of antibiotics from the first day of disease.
13. History/suspicion of oncology of any localization (except for benign neoplasms).
14. Exacerbation or decompensation of chronic diseases (diabetes mellitus, bronchial asthma, chronic bronchitis, chronic obstructive pulmonary disease, cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, malformations of the respiratory and ENT organs, etc.) affecting the patient's ability to participate in the clinical trial.
15. Previously diagnosed immunodeficiency of any etiology.
16. Unstable angina or myocardial infarction during the last 6 months.
17. Class III and IV chronic heart failure (according to the classification of the New York Heart Association, 1964).
18. History of chronic kidney disease (classes C3-5 A3).
19. History of liver failure (class C according to Child-Pugh).
20. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
21. Pregnancy, breast-feeding, and childbirth less than 3 months before inclusion in the trial.
22. Hypersensitivity to any component of the medicines used in the treatment.
23. Patients who used medications listed under "Prohibited Concomitant Treatment" within 1 month prior to inclusion in the trial or need medications prohibited for use in the trial.
24. Patients who, from the investigator's point of view, will not comply with the observation requirements during the trial or follow the procedure for taking the test drugs.
25. History of mental illness, alcoholism, drug abuse, which, from the investigator's point of view, will prevent the patient from following the trial procedures.
26. Participation in other clinical trials within 3 months prior to inclusion in this trial.
27. Patient is related to on-site research personnel directly involved in the trial, or is the immediate family member of the investigator. 'Immediate family members' mean spouses, parents, children, or siblings, whether related or adopted.
28. Patient is employed by OOO "NPF "MATERIA MEDICA HOLDING", i.e., is an employee of the company, a temporary contract employee, or a designated official responsible for conducting the trial or their immediate family member.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with improvement of acute rhinosinusitis symptoms on day 4 | On 4 day
  Improvement of symptoms is defined as symptom score less than or equal to 1 (i.e., mild symptoms or no symptoms) for all five main symptoms (rhinorrhea / anterior nasal discharge, postnasal drip, nasal congestion, headache, facial pain/pressure) with 2 consecutive 12-hour estimates.

SECONDARY OUTCOMES:
Percentage of patients with improvement of acute rhinosinusitis symptoms on day 7 | On 7 day of observation
  Improvement of symptoms is defined as symptom score less than or equal to 1 (i.e., mild symptoms or no symptoms) for all five main symptoms (rhinorrhea / anterior nasal discharge, postnasal drip, nasal congestion, headache, facial pain/pressure) with 2 consecutive 12-hour estimates.
Change in SNOT-22 total score | On days 1, 4 and 7
  Change in the Sino-Nasal Outcome Test (SNOT-22) total score from baseline to days 4 and 7 of observation. 22 symptoms are assessed. Symptom severity is rated on a scale of 0 to 5 (0 - no problem, 1 - very mild problem, 2 - mild or slight problem, 3 - moderate problem, 4 - severe problem, 5 - as bad as it gets). The maximum SNOT-22 score is 110.
Change in MSS total score | From day 1 to day 14
  Based on patient dairy. Change in MSS total score daily from baseline to day 14 of observation. Five main symptoms are assessed: runny nose/anterior nasal discharge, postnasal drip (need to cough mucus from the throat), nasal congestion, headache, facial pain/heaviness). The severity of symptoms is assessed in points from 0 to 3 (0 - none, 1 - mild, 2 - moderate, 3 - severe). The maximum total MSS score is 15 points. The total MSS score should not be less than 8 and not more than 12 points (inclusion criterion).
Change in the SNOT-22 nasal domain score | On days 1, 4 and 7
  Change in the SNOT-22 nasal domain score from baseline to days 4 and 7 of observation.
Percentage of patients with worsening of rhinosinusitis requiring systemic/topical antibiotics | On 14 day
  Percentage of patients with worsening of rhinosinusitis requiring systemic/topical antibiotics. Based on medical records.
Proportion of patients hospitalized due to worsening rhinosinusitis | On 14 day
  Proportion of patients hospitalized due to worsening rhinosinusitis. Based on medical records.
Percentage of patients with prolonged rhinosinusitis | On 14 day
  The percentage of patients with prolonged rhinosinusitis (main symptoms of the disease persisting for more than 7 days, progression of symptoms). Prolonged rhinosinusitis is defined as the persistence of the main symptoms of the disease, the progression of symptoms for more than 7 days, namely, the presence of the MSS symptoms rated as 2 or more points for one or more symptoms.
Number of Participants With Adverse Events (AEs) | From day 1 to day 14
  Presence and nature of adverse events during therapy. Registration of AEs begins after the first dose of the study drug, continues throughout the entire period of study therapy, and also for 24 hours after the last dose of the study drug. Based on medical records.
Severity of AEs | From day 1 to day 6
  The intensity (severity) of adverse events. Based on medical records.
Causal Relationship of AEs to the Sudy Drug | From day 1 to day 6
  The causal relationship to the study drug of adverse events. Based on medical records.
Outcome of AEs | From day 1 to day 6
  The outcome of adverse events. Based on medical records.
Changes in Vital Signs (Blood Pressure) | On days 1, 4 and 7
  Blood Pressure measured in mm Hg. Based on medical records.
Changes in Vital Signs (Heart Rate) | On days 1, 4 and 7
  Pulse Rate measured in beats per minute. Based on medical records.
Changes in Vital Signs (Breathing Rate) | On days 1, 4 and 7
  Respiratory Rate measured in breaths per minute. Based on medical records.

CONTACTS AND LOCATIONS:
Locations (39):
- Russia (39):
  - Aramil city hospital, Aramil
  - Gatchina Clinical Interdistrict Hospital, Gatchina
  - Baltic Federal University named after Immanuel Kant, Kaliningrad
  - Kazan State Medical University/Department of Infectious Diseases, Kazan'
  - Kuban State Medical University/Department of Infectious Diseases and Phthisiopulmonology, Krasnodar
  - First Moscow State Medical University named after I.M. Sechenov/Department of Ear, Nose and Throat Diseases, Moscow
  - National Medical Research Center of Otolaryngology, Moscow
  - Russian University of Medicine/Department of Otolaryngology, Moscow
  - Moscow Regional Research Clinical Institute named after M.F. Vladimirsky, Moscow
  - LLC "Persona Group of Companies", Nizhny Novgorod
  - Novosibirsk State Medical University/Department of Otolaryngology, Novosibirsk
  - LLC "Clinical and Diagnostic Center "Mediclinic", Penza
  - LLC "Professor's Clinic", Perm
  - Rostov Central District Hospital, Rostov
  - LLC "Otolaryngology Consultation Center", Rostov-on-Don
  - Rostov-on-Don City Hospital of Emergency Medical Care, Rostov-on-Don
  - North-West State Medical University named after I.I. Mechnikov/Department of Otolaryngology, Saint Petersburg
  - St. Petersburg Research Institute of Phthisiopulmonology, Saint Petersburg
  - City Polyclinic # 44, Saint Petersburg
  - LLC "Energy of Health", Saint Petersburg
  - LLC "Medical center "Reavita Med SPb", Saint Petersburg
  - LLC "Medical services", Saint Petersburg
  - LLC "Zvezdnaya Clinic", Saint Petersburg
  - First Saint Petersburg State Medical University named after I.P. Pavlov/Department of Otolaryngology with clinic, Saint Petersburg
  - City Polyclinic # 34, Saint Petersburg
  - Institute of Experimental Medicine, Saint Petersburg
  - City Polyclinic # 106, Saint Petersburg
  - City Pokrovskaya Hospital, Saint Petersburg
  - LLC "Meili", Saint Petersburg
  - Medical University "Reaviz", Samara
  - Samara State Medical University/Department of Otolaryngology, Samara
  - Saratov State Medical University named after V.I. Razumovsky/Department of Faculty Therapy, Saratov
  - LLC "Uromed", Smolensk
  - LLC "Scientific Medical Center of General Therapy and Pharmacology", Stavropol
  - Bashkir State Medical University/Department of Internal Medicine, Ufa
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - Clinical Hospital # 2, Yaroslavl
  - LLC "Medical center for diagnostics and prevention plus", Yaroslavl
  - Ural State Medical University/Department of Surgical Dentistry, Otorhinolaryngology and Maxillofacial Surgery, Yekaterinburg